CLINICAL TRIAL: NCT05134428
Title: Open-label, Dose Ranging, Multi-Centre, Prospective First in Human Study to Assess the Safety of the ADAM System
Brief Title: A First in Human Study, Evaluating the Safety and Efficacy of ADAM™ 1.0
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Contraline, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: ADM-012
Record Dates: First submitted 2021-11-13; First posted 2021-11-26 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Male Contraception; Healthy Male Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- ADAM Cohort 1 (Experimental): The first 5 subjects will be reviewed for safety by a Data Safety Monitoring Board (DSMB) at 30 days post-implantation. The 5 subjects will then be followed up to 24 months or until their semen analyses is ≥ 15 million sperm/mL.
  Interventions: Device: ADAM System
- ADAM Cohort 2 (Experimental): An additional 13 subjects will be enrolled and implanted with ADAM. They will be followed up to 24 months or until or until their semen analyses is ≥ 15 million sperm/mL.
  Interventions: Device: ADAM System
- ADAM Cohort 3 (Experimental): An additional 4 subjects will be enrolled and implanted with ADAM. They will be followed up to 24 months or until or until their semen analyses is ≥ 15 million sperm/mL.
  Interventions: Device: ADAM System
- ADAM Cohort 4 (Experimental): An additional 3 subjects will be enrolled and implanted with ADAM. They will be followed up to 24 months or until or until their semen analyses is ≥ 15 million sperm/mL.
  Interventions: Device: ADAM System

INTERVENTIONS:
Device: ADAM System — The ADAM System consists of an injectable hydrogel and delivery apparatus that is intended to provide long-lasting, non-permanent vasal occlusion for men, resulting in azoospermia. ADAM is designed to be inserted into the vasa deferentia through a minimally invasive procedure, similar to the no-scalpel vasectomy.

SUMMARY:
This study will evaluate the safety and feasibility of the ADAM System for implantation into the vas deferens in 25 healthy males at 3 sites. This is a prospective, non-randomized, open label interventional trial.

DETAILED DESCRIPTION:
The ADAM System consists of the ADAM Hydrogel and the ADAM Injector. The ADAM Hydrogel is a proprietary, injectable, co-polymer hydrogel designed to provide long-lasting, non-permanent vasal occlusion for men. The ADAM Injector automates the dose and speed at which the ADAM Hydrogel is delivered into the vas deferens. The vas deferens may be accessed using a minimally invasive no-scalpel technique. Once inserted into the lumen of the vas deferens, the hydrogel prevents sperm transport from the epididymis into the ejaculate.

Subjects will be followed up to 24 months or until semen analysis is ≥ 15 million sperm/mLA second semen analysis may be required to confirm sperm concentration, this is to be requested at the discretion of the study investigator, the second sample must be collected ≥2 days and ≤10 days of the first).

The 25 subjects will be enrolled as follows:

A minimum of 3 and up to 13 in each cohort. The Cohorts will enroll in parallel.

The DSMB will meet at various timepoints during the study to review the safety data from the subjects (up to the 30-day post implant visit), e.g. after the first 4-5 subjects in any given cohort. Appropriate action will be taken if any related event is observed.

Pre-procedure, the subject will provide two separate semen samples for lab analysis, the results of which will be averaged. The duration between collection of both specimens will be ≥2 days and ≤7 days. This will determine baseline sperm count and eligibility for enrolment.

All subjects who demonstrate azoospermia or virtual azoospermia post-procedure will be followed until the semen analysis at any designated timepoint/visit demonstrates a sperm concentration ≥ 15 million sperm/mLthe lower 5% reference limit according to the WHO Laboratory Manual for the Examination and Processing of Human Semen). The subject may subsequently undergo a second lab semen analysis within 2-10 days to confirm the sperm concentration (decided at the discretion of the study investigator). If the subject's sperm concentration is still not conclusive after the second analysis, they will remain on trial until conclusive results are achieved. The subject's participation in the study will end once their semen analysis demonstrates ≥ 15 million sperm/mL or at 24 months after ADAM implantation, whichever is sooner. Subjects who do not achieve azoospermia by month 12 will be exited from the study. For clarity, subjects will remain in the study for a minimum of 12 months whether or not they achieve azoospermia or until resolution of any adverse event. Subjects whose participation in the study ends will be offered a vasectomy.

An alternative form of contraception will be required for the duration of the study regardless of whether the subject demonstrates azoospermia during the course of the study.

Lab Samples: All lab samples will be destroyed as per the local lab standard policy. The samples will not be retained for any further analysis or research.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is male
2. Subject is 25 to 65 years of age
3. Subject has a normal semen analysis (≥ 15 million sperm/mL, ≥40% total motility) defined by the WHO Laboratory Manual for the Examination and Processing of Human Semen (5th Edition), based on the average of two semen samples ≥2 days and ≤7 days apart
4. Subject is suitable to undergo a vasectomy as a long-term form of contraception
5. Subject is legally competent
6. In the opinion of the Investigator, the subject is willing and able to comply with the protocol, return for all follow-up visits and complete all protocol assessments, which includes providing recurring semen samples
7. Subject agrees to use an alternative method of contraception with any female partner of reproductive age during the course of the study treatment until study exit occurs
8. Subject is willing to accept an unknown risk of conceiving a pregnancy during the duration of the study.
9. The subject has been informed of the nature of the study, agrees to its provisions, and has willingly provided written informed consent, approved by the appropriate Human Research Ethics Committee (HREC)

Exclusion Criteria:

* Potential subjects will be excluded if ANY of the following criteria apply:

  1. Subject is participating in another interventional clinical trial currently or within the past 3 months from the time of screening
  2. Subject has history of prior hormonal therapy use (e.g., androgenic steroids, GnRH agonists and antagonists) within the past 6 months
  3. Subject on exam has any of the following: vas not present, abnormal scrotum, large varicocele, hydrocele, filariasis or elephantiasis of scrotum, or intrascrotal mass that would make the subject not suitable for the study
  4. Subject has allergic reaction to polyethylene glycol (PEG) containing products or has had a prior severe allergic response to injectable or implantable devices
  5. Subject has local genital infections such as balanitis, scrotal skin infection, epididymitis, or orchitis, or tender (inflamed) tip of the penis, but may be admitted after resolution of an acute infection
  6. Subject has current coagulopathy or other bleeding disorders
  7. Subject currently taking or planning to take any type of systemic medication which could affect sperm count or ejaculation (e.g., anabolic steroids, chemotherapy, alpha blocker)
  8. Subject had a previous successful or unsuccessful vasectomy or vasectomy reversal
  9. Subject has any clinically significant abnormal findings or other findings identified by Investigator that would exclude the subject.

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 30 Days
  The primary endpoint is the number of all treatment-emergent adverse events

SECONDARY OUTCOMES:
Serious AEs | 30 Days
  Number and percentage of subjects experiencing procedure and device-related serious adverse events at 30 days
Adverse Events of Interest | 3 years
  Number and percentage of subjects experiencing an adverse event of interest during the study
Azoospermia | 3 years
  Percentage of subjects achieving absolute azoospermia, defined as a zero sperm count, and percentage of subjects achieving virtual azoospermia, defined as a sperm count of ≤100,000 per mL and 0% motility

CONTACTS AND LOCATIONS:
Overall Officials: Alex Pastuszak, MD, PhD, Study Director — Contraline, Inc; Nathan Lawrentschuk, MB, BS, PhD, FRACS, Principal Investigator — Epworth Healthcare
Locations (3):
- Australia (3):
  - South Coast Urology, Wollongong, New South Wales
  - AndroUrology, Brisbane, Queensland
  - Epworth HealthCare, East Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No